CLINICAL TRIAL: NCT06064019
Title: Evaluation of the Clinical Utility of a New Diagnostic Support Tool, Based on Electrical Impedance Spectroscopy (NEVISENSE), for Keratinocyte Skin Cancer
Brief Title: Evaluation of Nevisense as Support Tool for the Diagnose of Keratinocyte Skin Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SciBase AB (Other)
Responsible Party: Principal Investigator, Thomas Dirschka, Prof Dr, CentroDerm GmbH
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EIS-KC001
Record Dates: First submitted 2023-09-11; First posted 2023-10-03 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Keratinocyte Skin Cancer
Keywords: Electrical Impedance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Nevisense (Other): This will be a prospective investigator-initiated study to evaluate the accuracy of Nevisense for KC. First evaluation steps include dermatologist's clinical examination (visual inspection) and videodermoscopy. In those cases where the routine diagnostic procedures given above identify any suspicion of a KC, a Nevisense measurement is to be conducted after examination of inclusion and exclusion criteria. Thereafter, surgical excision and histopathologic examination follow.
  All skin lesions with a suspicion of BCC, iSCC, BD or AK and destined for excision or biopsy for further histopathological analysis will be considered for inclusion in the study. A maximum of three lesions per patient will be allowed for the study. The study aims to enrol 250 lesions in total.
  Interventions: Device: Nevisense

INTERVENTIONS:
Device: Nevisense — The Nevisense system is based on Electrical Impedance Spectroscopy (EIS). EIS is a measure of the overall resistance within a skin tissue, at alternating currents of various frequencies. Since skin tissues have different electrical properties depending on cell structure and medical conditions, the resulting electrical impedance spectra will reflect the properties of the skin tissue.

SUMMARY:
This is a prospective study to assess efficacy of the Nevisense device in identifying keratinocyte skin cancer (KC) in patients suspected of having skin cancer based on the initial physician's assessment.

All skin lesions with a suspicion of Basal cell carcinoma (BCC), Invasive Squamos cell Carcinoma (iSCC), Bowen's disease (BD) or actinic keratosis (AK) and destined for excision or biopsy for further histopathological analysis will be considered for inclusion in the study.

ELIGIBILITY:
Inclusion Criteria:

* All male or female patients of any ethnicity, ≥ 18 years with skin lesions of a clinical uncertain diagnosis suspicious for KC (such as BCC, iSCC, BD or AK)

Exclusion Criteria:

* Metastases of recurrent lesions
* Lesion located on acral skin, e.g. sole or palm
* Lesion located on areas of scars, crusts, psoriasis or similar skin conditions
* Lesion on hair-covered areas, e.g. scalp, beards, moustaches
* Lesion located on genitalia
* Lesion located in an area that has been previously biopsied or subjected to any kind of surgical intervention or traumatized
* Lesion located on mucosal surfaces
* Lesion with foreign matter, e.g. tattoo or splinter
* Lesion and / or reference located on acute sunburn
* Skin surface not measurable, e.g. lesion on a stalk
* Skin surface not accessible, e.g. inside ears, under nails

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-07-13 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Nevisense Sensitivity and Specificity | 1 year
  This study has two primary endpoints:
  1. Sensitivity ≥ 0.90
  2. Sensitivity + Specificity > 1.0
  Sensitivity is the proportion of correctly identified cases of KC. Specificity is the proportion of correctly identified cases of non-KC

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Dirschka, Prof. Dr. med., Principal Investigator — CentroDerm GmbH
Locations (1):
- CentroDerm, Wuppertal, Germany